CLINICAL TRIAL: NCT04912258
Title: Trans-arterial Chemoembolization With Irinotecan Drug-eluting Beads Before Liver Surgery for Patients With Primary Unresectable Colorectal Liver Metastasis: A Randomized Control Trial
Brief Title: Preoperative Irinotecan Drug-eluting Beads for Patients With Unresectable Colorectal Liver Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIDUC
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): DEB-TACE before liver surgery
  Interventions: Drug: Trans arterial chemoembolization with Irinotecan Drug-eluting Beads
- Arm B (No Intervention): direct liver surgery

INTERVENTIONS:
Drug: Trans arterial chemoembolization with Irinotecan Drug-eluting Beads — preoperative chemoembolization with Irinotecan Drug-eluting Beads
  Other Names: Irinotecan Drug-eluting Beads
  Arms: Arm A

SUMMARY:
Trans arterial chemoembolization using Irinotecan Drug-eluting Beads before liver surgery for patients with primarily unresectable colorectal liver metastasis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histologically proven colorectal liver metastasis；
* With liver-dominant disease；
* Primarily evaluated as potentially resectable and conversed successfully
* Adequate hematologic function: absolute neutrophil count (ANC)≥1.5×109/l, platelets≥75×109/l, and international normalized ratio (INR) ≤1.3 (within 1 week prior to randomization)
* Adequate liver and renal function: total bilirubin ≤2.0 mg/dl, alanine aminotransferase, aspartate aminotransferase ≤ 5x upper limit of normal, and albumin≥2.5 g/dl, serum creatinine≤2.0 mg/dl (within 1 week prior to randomization);
* Written informed consent for participation in the trial.

Exclusion Criteria:

* Primarily evaluated as resectable
* Failed to converse
* Patients with known hypersensitivity reactions to any of the components of the study treatments.
* Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
* Other previous malignancy within 5 years
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
liver relapse-free survival | 6 months
  from liver surgery to liver relapse

SECONDARY OUTCOMES:
relapse-free survival | 6 months
overall survival | 12 months
response rate | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided